CLINICAL TRIAL: NCT05769725
Title: A Study to Evaluate Serplulimab in Combination With Docetaxel +S-1 VS. Docetaxel +S-1 as Adjuvant Treatment Therapy in Stage IIIc Gastric Cancer(PD-L1 + / MSI-H / EBV +/dMMR)
Brief Title: A Study to Evaluate Serplulimab in Combination With Docetaxel +S-1 VS. Docetaxel +S-1 as Adjuvant Treatment Therapy in Stage IIIc Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0001
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Serplulimab,Gastric Cancer, Adjuvant Therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulimab in Combination With Docetaxel +S-1 (Experimental)
  Interventions: Drug: Serplulimab; Drug: Docetaxel; Drug: S1
- Docetaxel +S-1 (Placebo Comparator)
  Interventions: Drug: Docetaxel; Drug: S1

INTERVENTIONS:
Drug: Serplulimab — Serplulimab, 4.5mg/kg solution intravenously for 30 min in first day every 3 weeks. Repeated every 21 days. 21 days for a cycle.
  Other Names: HLX10
  Arms: Serplulimab in Combination With Docetaxel +S-1
Drug: Docetaxel — 40 mg/m^2 solution intravenously for 1 hour in first day every 3 weeks. Repeated every 21 days, 21 days for a cycle, from second cycle to seventh cycle.
Drug: S1 — Tegafur-gimeracil-oteracil potassium: 50mg bid orally in 14 days, followed by 7 days off. Rrepeated every 21 days. 21 days for a cycle.

SUMMARY:
To evaluate the efficacy and safety of Serplulimab in Combination With Docetaxel +S-1 vs. Docetaxel +S-1 as Adjuvant Treatment Therapy in Stage IIIc Gastric Cancer (PD-L1 + / MSI-H / EBV +/dMMR) . Secondary study objective: To observe and evaluate the overall survival and adverse events of Serplulimab in Combination With Docetaxel +S-1 vs. Docetaxel +S-1 as Adjuvant Treatment Therapy in Stage IIIc Gastric Cancer (PD-L1+ / MSI-H / EBV +/dMMR). To evaluate the safety of Serplulimab in Combination With Docetaxel +S-1 vs. Docetaxel +S-1 as Adjuvant Treatment Therapy in Stage IIIc Gastric Cancer (PD-L1 + / MSI-H / EBV +/dMMR). To explore the incidence of PD-L1 + / MSI-H / EBV + /dMMR in stage IIIc gastric cancer. To explore the correlation of PD-L1 + / MSI-H / EBV + /dMMR in stage IIIc gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patients voluntarily joined the study and signed the informed consent; ≥ 18 years old, ≤ 75 years old, both male and female; Stage III gastric cancer confirmed by pathology, ECoG score: 0-1 Detection of biomarkers in postoperative gastric cancer samples suggests that: PD-L1 + CPS ≥ 5 / MSI-H + / EBV+/dMMR No preoperative anti-tumor treatment for gastric cancer, including chemotherapy and local treatment During the study treatment period and within 3 months after the end of the study treatment period, a medically recognized contraceptive measure (such as IUD, contraceptive pill or condom) should be used for the female patients of non-surgical sterilization or childbearing age; the serum or urine HCG test of the female patients of non-surgical sterilization must be negative within 72 hours before the study group; and the hCG test must be non lactation; for the male patients Sex, should be surgical sterilization, or agree to use appropriate methods of contraception during the trial and within 3 months after the last administration of the test drug.

The baseline blood routine and biochemical indexes of the selected patients should meet the following standards:

A. hemoglobin ≥ 90g / L

B. absolute neutrophil count ≥ 1.5 × 10 ^ 9 / L

C. platelet count ≥ 100 × 10 ^ 9 / L

D. ASTor ALT ≤ 2.5 ULN

E. Alkaline phosphatase (ALP)≤ 2.5×ULN

TSH ≤ 1 ULN (if abnormal, T3 and T4 levels should be examined at the same time, if T3 and T4 levels are normal, they can be included in the group);

Exclusion Criteria:

* Pregnant or lactating women; Women of childbearing age were positive in the baseline pregnancy test; Distant metastasis was diagnosed by CT /MR/ EUS. Received previous anti-tumor treatment, including chemotherapy, radiotherapy or immunotherapy; Have other malignant tumors in the past 5 years (except basal cell or squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ or breast cancer); Uncontrollable pleural effusion, pericardial effusion or ascites; Severe cardiovascular diseases such as symptomatic coronary heart disease, congestive heart failure ≥ level II, uncontrolled arrhythmia and myocardial infarction within 12 months before admission; With gastroduodenal obstruction/bleeding, digestive dysfunction or malabsorption syndrome Complicated with severe uncontrolled concurrent infection or other serious uncontrolled concomitant diseases, moderate or severe renal injury; Allergic reaction to the drugs used in this study; Steroid or other systemic immunosuppressive therapy was used 14 days before admission; Patients who received study drug treatment within 4 weeks before enrollment (participate in other clinical trials).

Active autoimmune diseases (including but not limited to: uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchodilator treatment). Subjects with hypothyroidism requiring only hormone replacement therapy and skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia) can be selected.

History of primary immunodeficiency. Immunosuppressive drugs were used within 4 weeks prior to the first dose of study treatment, excluding local or physiological doses of systemic glucocorticoids (i.e. no more than 10mg / day of prednisone or other glucocorticoids of equivalent dose) by nasal spray, inhalation or other routes, or hormones used to prevent allergy of contrast agents.

Receive live attenuated vaccine within 4 weeks before the first dose of study treatment or during the study period.

Active tuberculosis is known. We have known the history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.

HIV antibody positive, active hepatitis B or C (hepatitis B: HBsAg positive and HBV DNA ≥ 10 ⁴ copies / ml; hepatitis C: HCV antibody and HCV-RNA positive, requiring antiviral treatment at the same time);.

Other factors that may affect the safety or test compliance of the subjects according to the judgment of the researchers. For example, serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, or other family or social factors, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 1 years
  disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Zizhen, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided